CLINICAL TRIAL: NCT04965987
Title: A Phase I, Double-Blind, Pilot Study of Oxaloacetate in Myasthenia Gravis
Brief Title: Oxaloacetate in Myasthenia Gravis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Terra Biological LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MG OAA
Record Dates: First submitted 2021-06-10; First posted 2021-07-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Oxaloacetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxaloacetate (Active Comparator): Oxaloacetate (OAA) is a four-carbon molecule involved in many metabolic pathways, including gluconeogenesis, citric acid cycle, glyoxylate cycle, urea cycle, and amino acid metabolism. In the glyoxylate and citric acid cycles, oxaloacetate is formed as the result of the catalysis by malate dehydrogenase.
  Subjects will take 1000mg OAA BID for 8 weeks.
  Interventions: Drug: Oxaloacetate
- Placebo (Placebo Comparator): Subjects will take 1000mg Placebo BID for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxaloacetate — Oxaloacetate (OAA) is a four-carbon molecule involved in many metabolic pathways, including gluconeogenesis, citric acid cycle, glyoxylate cycle, urea cycle, and amino acid metabolism. In the glyoxylate and citric acid cycles, oxaloacetate is formed as the result of the catalysis by malate dehydrogenase. In this reaction, the hydrogen atoms from malate are transferred to NAD+, forming NADH, H+ and oxaloacetate. Oxaloacetate can be converted to citrate with the addition of acetyl-CoA by the enzyme citrate synthase. Oxaloacetate is a critical component in the production of ATP and must be constantly regenerated in order for the citric acid cycle and the electron transport chain to continue
  Other Names: CRONaxal
  Arms: Oxaloacetate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase 1 clinical trial studying whether or not oxaloacetate has a positive effect on patients with Myasthenia Gravis. Patients will be assigned to one of three cohorts which will determine the dose of oxaloacetate they will be given. Subjects will take the study drug for 4 weeks and be on placebo for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 and older.
2. Patients must have prior or current documentation of MGFA MG grades 2, 3, or 4A generalized MG, according to the MGFA classification system. These grades correspond to mild (2), moderate (3), and severe (4).
3. A total MG-ADL score of greater than 3 at Screening and Baseline with no more than 50% of the total score being due to ocular symptoms.
4. Patient's signs and symptoms should not be better explained by another disease process.
5. Patients must be willing to complete the study and return for follow-up visits.
6. Patients must be willing to give written informed consent before participating in this study. A copy of the signed consent must be kept in the patient's medical record.
7. Patients can be on the following drugs as long as there has been no dose change for 60 days: azathioprine, cyclosporine, cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate, IVIg or other immunosuppressive drugs.
8. Patients can be on prednisone as long as there has been no dose change for 30 days.
9. No planned changes in MG medications during the study

Exclusion Criteria:

1. MGFA grade V within 6 months of screening.
2. A history of chronic degenerative, severe psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue.
3. Other major chronic or debilitating illnesses within six months prior to study entry.
4. Female patients who are premenopausal and are: (a) pregnant on the basis of a serum pregnancy test, (b) breast-feeding, or (c) not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures).
5. Thymectomy in the previous three months.
6. History of severe reactions to OAA
7. Participation in a research study within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Frequency and Severity of Adverse Events) | At weeks 2, 4, 6, 8, 10, and 12
  The primary endpoint of safety will be reported as counts of subjects experiencing adverse events events (including abnormal laboratory results and vital signs). Measures of safety will be reported for the last visit observed for each participant.

SECONDARY OUTCOMES:
Myasthenia Gravis-specific Activities of Daily Living Scale (MG-ADL) Score | Change from Week 4 to Week 8
  Myasthenia Gravis-specific Activities of Daily Living scale (MG-ADL): Composite measure of scores from measurement scales. The MG-ADL has a scale of 0 - 24 with 0 being the lowest (no symptoms) and 24 being the highest (most severe symptoms. The MG-ADL is a staff-administered, patient-reported questionnaire that measures 8 commons symptoms of myasthenia gravis and grades them on a scale of 0 - 3.
Quantitative Myasthenia Gravis (QMG) Score | Change from Week 4 to Week 8
  The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The scale is from 0 - 3 for each item, with 0 meaning normal and 3 is severe. Total score can range from 0 to 39.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States